CLINICAL TRIAL: NCT01692873
Title: Research for Prognostic and Predictive Biomarkers of Therapeutic Response in Pancreatic Tumors - PACAomics / IPC 2011-004
Brief Title: Prognostic and Predictive Biomarkers of Therapeutic Response in Pancreatic Tumors
Acronym: PACAomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PACAomics / IPC 2011-004
Record Dates: First submitted 2012-09-14; First posted 2012-09-25 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Tumor
Keywords: pancreatic tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- suspected pancreatic tumor (Experimental): Realization of pancreatic tumor biopsy and blood samples
  Interventions: Procedure: suspected pancreatic tumor

INTERVENTIONS:
Procedure: suspected pancreatic tumor — Realization of pancreatic surgery to obtain tumor biopsy and blood samples to realize biomarkers analyses.

SUMMARY:
Pancreatic cancer is among the most serious human neoplasia and the most difficult to treat.

Most patients present at diagnosis a non resectable, locally advanced or metastatic disease, with a median survival of 12 month.

The aim of this study is the identification of diagnosis biomarkers, predictive of the therapeutic response.

This project investigate the use of molecular analyses applied to pancreatic tumor cells collected by microbiopsy under ultrasound-endoscopy, and blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of pancreatic adenocarcinoma
* Patient > 18 years old
* Social Security affiliation
* Signed informed consent

Exclusion Criteria:

* Patient in emergency situation
* Major person being the object of a legal protective measure or unable to express its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2012-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers | within twenty four hours
  Genomics, transcriptomics and proteomics analyses to determine presence or absence of biomarkers

SECONDARY OUTCOMES:
Histology | within twenty four hours
  To determine the histologic characteristics of the pancreatic tumor

CONTACTS AND LOCATIONS:
Overall Officials: Marine GILABERT, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Marine GILABERT, MD, Marseille, France

REFERENCES:
- [Derived] Fraunhoffer NA, Abuelafia AM, Chanez B, Bigonnet M, Gayet O, Roques J, Chuluyan E, Dusetti N, Iovanna J. Inhibition of glucuronidation in pancreatic cancer improves gemcitabine anticancer activity. Cancer Commun (Lond). 2022 Nov;42(11):1212-1216. doi: 10.1002/cac2.12365. Epub 2022 Sep 30. No abstract available. PMID 36178036
- [Derived] Fraunhoffer NA, Abuelafia AM, Dusetti N, Iovanna J. Limitation and challenges in using pancreatic cancer-derived organoids as a preclinical tool. Cancer Commun (Lond). 2022 Oct;42(10):1028-1031. doi: 10.1002/cac2.12335. Epub 2022 Jul 18. No abstract available. PMID 35848462
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr/